CLINICAL TRIAL: NCT07219381
Title: The Impact of Holistic Medicine Treatment for Bachelorettes Residing on Tribal Lands or in the State of Alaska Living With Uterine Fibroids-1St Diagnosis, Uterine Fibroids Affecting Pregnancy, or Uterine Fibroid Degenerated
Brief Title: Holistic Medicine Treatment of Uterine Fibroids-Adults
Acronym: HMTXUFAdult
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Virtual Tribunal Monastery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RYXWWMJUDPM6-Bachelorettes
Record Dates: First submitted 2025-10-08; First posted 2025-10-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Uterine Fibroids - 1St Diagnosis; Uterine Fibroids Affecting Pregnancy; Uterine Fibroid Degenerated
MeSH Terms: interventions — Holistic Health

STUDY DESIGN:
Intervention Model Description: Holistic Medicine, also known as Holistic Education, represents a nonclinical approach to healing, recovery and wellness. It focuses on nurturing the whole person-mind, body, and spirit-to achieve optimal well-being. Other names for this intervention include Nonclinical Variables and Adult Education.
  The Patient-Centered Medical Home (PCMH) model plays a crucial role in delivering holistic care. PCMH provides individualized care, patient engagement, and comprehensive care coordination within a single practice. The ultimate goal is to improve quality of life through prevention education, treatment, and rehabilitation programs tailored to individual patient needs.
  Holistic Medicine (Holistic Education) emphasizes patient self-help and self-care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resource Utilization Group (RUG) (Experimental): nonclinical variables
  Interventions: Behavioral: Holistic Medicine (HM)

INTERVENTIONS:
Behavioral: Holistic Medicine (HM) — With informed consent the participant act as a partner to their health and acknowledges responsibility for self-help or self-care directed activities in a non-clinical setting. Transcendence in research involves actively exploring the best possible options or resources for a resolution or self-determination or hypotheses. To reinforce healthy activities, periodic forecast consist of one or more of the following variables: pastoral counseling, lectures, group discussions, sound therapy, team building exercises, faith-based initiatives, outdoor exercise, walking group, support group, supportive care, cooking class, critical thinking questioning and self-assessment tests. Adult content variables are classified under gender-specific care Respite ( i.e. watch party, gaming, music therapy, interactive Spiritual story, clothing model therapy, portable foot spa and portable foot massage) TO (Time-Out).
  Other Names: Holistic Education; Transcendence Research; Adult Education

SUMMARY:
This clinical trial aims to evaluate the efficacy of holistic medicine treatments for unmarried women ("Bachelorettes") residing on U.S. Tribal Lands or in the State of Alaska who have been clinically diagnosed with uterine fibroids. The study will assess both primary and secondary outcomes, while accounting for socioeconomic and cultural factors that may influence treatment efficacy and data validity. The research acknowledges the unique sociocultural and economic contexts of Tribal communities and aims to contribute to equitable healthcare research practices, with particular attention to urban poverty, unmarried status, and substance-free lifestyle factors.

DETAILED DESCRIPTION:
OBJECTIVES:

To evaluate the clinical efficacy of holistic medicine treatments for uterine fibroids among unmarried women on Tribal Lands or in the State of Alaska, with focus on urban and economically disadvantaged populations.

To assess the influence of socioeconomic factors including urban poverty, marital status, and substance-free lifestyle choices on treatment outcomes.

To identify barriers to participation and data validity arising from systemic inequities affecting Tribal communities and urban populations experiencing poverty.

ELIGIBILITY:
Inclusion Criteria: To join this study, you must meet these simple requirements:

* Be a Bachelorette Alaska Medicaid recipient age 21 years old and older.
* Have been told by a doctor that you have uterine fibroids (non-cancerous growths in your uterus).
* Live on Tribal Lands or anywhere in the State of Alaska,
* Be willing to try natural, nonclinical holistic treatments alongside regular clinical medical care.
* Acknowledge smoke-free, drug-free, and alcohol-free church policy
* Must have access to the internet, Holy Bible (KJV) and a portable fetal Doppler to listen to and monitor uterine fibroid heart rate in spiritual mysteries.
* Religious or spiritual belief in prayer meditation for faith-based healing.
* Must agree to medical ethical standards in Greek text pertaining to the Hippocratic Oath.
* Due to a new tool in the Toolkit: DOGS HELP TO DETECT COVID-19, a negative COVID-19 test may be required at any time whenever COVID-19 is suspected without remedy.

You May Still Qualify Even If:

* You haven't tried other treatments yet.
* You're currently receiving other fibroid treatments.
* You live in a remote area with limited healthcare access.
* You prefer natural or traditional healing approaches.
* You have concerns about surgery or medications.

Exclusion Criteria:

* Noncompliance to Inclusion Criteria.
* Married relationship status
* Gender conversion
* Repeat Offenders
* Ineligible for Alaska Medicaid
* Smokers, vapors, alcoholics, drug abusers.
* Non-Believers in Christian religious practices or prayer.
* Immobility
* Diseases without clinical diagnosis, medical treatment, and remedy.
* Uterine Fibroids premature removal by invasive/noninvasive surgery or Birth Control before climacteric.
* Unreported violence or abuse can inadvertently influence the validity of this study.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2029-01-19 (Estimated); Study Completion 2029-01-19 (Estimated)

PRIMARY OUTCOMES:
Holistic Medicine Qualitative Method | 1 year
  Qualitative data are not expressed numerically. Qualitative evaluation method summarize evidence from instructed methods of data collection relevant to socioeconomic factors, naturalistic observation, and existing records. Hierarchy scales of evaluation determine client wellness stages and identify areas requiring additional nonclinical variables for optimum wellness.

SECONDARY OUTCOMES:
Holistic Medicine Quantitative Method | 1 year
  Based on an average score total 1-100 point scale questionnaire, self-assessment, and/or critique forms will be used to measure socioeconomic factors as well as behaviors, impact, reaction, coping, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Jones, Study Chair — Humanitarian Veterans Association
Locations (1):
- Virtual Tribunal Monastery, Anchorage, Alaska, United States

REFERENCES:
- [Result] Jones G. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. Transcendence Research. 2025 December; 1(1).
- [Result] Jones G. Transcendence Research: Counterterrorism to Prevent Victimization. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. 2025 December; 1(2).
- [Result] Jones G. Transcendence Research: Holistic Healthcare for Social-Welfare Inequities Pursuant to Chronic Health Conditions. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. 2026 January; 2(1).
- See also: means-tested benefits — https://studentaid.gov/help/means-tested-benefits
- See also: doppler — https://www.webmd.com/baby/pregnancy-fetal-heart-monitoring#1-4
- See also: climacteric — https://dictionary.apa.org/climacteric
- See also: Liaison — https://djewss.my.canva.site/veterans-report-form
- See also: Greek Medicine — https://www.nlm.nih.gov/hmd/topics/greek-medicine/index.html
- See also: Virtual Tribunal Monastery Facility — https://virtualtribunalmonastery.vhx.tv/
- See also: A New Tool in the Toolkit: Dogs Help to Detect COVID-19 — https://www.cdcfoundation.org/stories/project-uses-dogs-detect-covid-19
- See also: Government Shutdown Clock — https://www.whitehouse.gov/government-shutdown-clock/